CLINICAL TRIAL: NCT06352827
Title: Guideline to Implementation: A Rapid Clinical Care Pathway to Care for Patients Affected by Chronic Constipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Eric Shah, Associate Professor of Internal Medicine, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM00228948; 1K23DK134752-01 (NIH)
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Constipation
Keywords: Questionnaires; Gastroenterology care
MeSH Terms: conditions — Constipation | interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: Participants will be enrolled in the observational intervention group first.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Observational Cohort (Other): This cohort will complete a baseline survey.
  Interventions: Behavioral: Survey

INTERVENTIONS:
Behavioral: Survey — All participants will complete a baseline survey and have medical information collected.

SUMMARY:
The study is being completed to test the pilot implementation of a rapid clinical care pathway for chronic constipation in the University of Michigan Gastroenterology clinic. This study will learn how often patients get better and how satisfied patients are with care decisions, when seen by a gastroenterologist for medical advice on constipation.

DETAILED DESCRIPTION:
Per the NIH requirements the study team added the following language and also updated the registration to be an interventional study. The study will enroll adult patients with chronic constipation prior to appointment with a gastroenterologist that have not received anorectal function testing or treatment in the past. The study team will assess patients' constipation symptoms and then monitor whether providers order anorectal function testing or treatment as a primary outcome. Source data will be derived from the medical record to provide quality assurance. The sample size is necessary to evaluate this outcome measure while accounting for missing data to address situations where variables are reported as missing, unavailable, non-reported, uninterpretable, or considered missing because of data inconsistency or out-of-range results. The statistical analysis plan will be descriptive with reporting of our binary primary endpoints given the nature of this being a pilot study.

Registration NCT07032376 (Implementation Phase) is part of this registration, "Guideline to Implementation: A Rapid Clinical Care Pathway to Care for Patients Affected by Chronic Constipation" (Observational Phase) NCT06352827.

ELIGIBILITY:
Inclusion Criteria Participants:

* Participant has Chronic constipation as a main symptom
* Participant is able to participate in pelvic floor physical therapy

Exclusion Criteria Participants:

* Participant has taken narcotic pain medication in the past 30 days
* Participant has been scheduled for a test called an anorectal manometry in the past
* Participant has been scheduled to see a pelvic floor physical therapist in the past
* Participant is pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2024-07-30 (Actual); Primary Completion 2025-08-08 (Actual); Study Completion 2025-08-08 (Actual)

PRIMARY OUTCOMES:
Percentage of encounters in which anorectal physiology testing is ordered or performed at the baseline routine-care gastroenterology office appointment | Day 1 (Baseline = initial appointment after consent)
  Fidelity to ordering pelvic floor diagnostics
Percentage of encounters in which pelvic floor physical therapy is ordered at the baseline routine-care gastroenterology office appointment | Day 1 (Baseline = initial appointment after consent)
  Fidelity to ordering pelvic floor treatment

CONTACTS AND LOCATIONS:
Overall Officials: Eric Shah, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-11-20): https://cdn.clinicaltrials.gov/large-docs/27/NCT06352827/ICF_000.pdf